CLINICAL TRIAL: NCT05755763
Title: Validity and Reliability of the Turkish St. Marks Incontinence Score
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Yasemin Ecem Temel Pekmez, Principal Investigator, Atlas University
Other Study IDs: YETPekmez
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Fecal Incontinence; Pelvic Floor Disorders
MeSH Terms: conditions — Fecal Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anal incontinence patients with St. Mark's Incontinence Score — The scale was applied to the patients who applied to our clinic with the diagnosis of anal incontinence.

SUMMARY:
For the Turkish validity and reliability study of St.Mark's (Vaizey) Incontinence Score, which consists of 7 questions, it will be applied to 65 people diagnosed with anal incontinence after it is translated by translation-retranslation method.

ELIGIBILITY:
Inclusion Criteria:

* people with the complatint of anal incontinence
* being volunteered to participate

Exclusion Criteria:

- having difficulties in understanding and speaking Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who were diagnosed with anal incontinence in our clinic will be included in the study. Persons who have difficulties in understanding and writing Turkish will be excluded from the study. Patients will fill out the St. Mark's Incontinence Score.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Turkish Validation and Reliability of St. Mark's Incontinence Score | 1 month
  St. Mark's Incontinence Score which shows the disease severity of anal incontinence patients and is used in the follow-up of their recovery status. The Turkish validity and reliability study of Mark's incontinence score will be conducted and it will be translated into Turkish.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Atakent University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided